CLINICAL TRIAL: NCT06938815
Title: A Novel Regimen for Treatment and Prevention of Post-Inflammatory Hyperpigmentation in Skin of Color
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Narrows Institute for Biomedical Research (Other)
Collaborators: L'Oreal (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1792718
Record Dates: First submitted 2025-04-02; First posted 2025-04-22 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-02

CONDITIONS: Post Inflammatory Hyperpigmentation
Keywords: skin of color; post inflammatory hyperpigmentation; skinceuticals
MeSH Terms: conditions — Hyperpigmentation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pigment Balancing Peel and Post Peel Regimen (Experimental): Discoloration Defense Serum: Applied twice daily (morning and night) LHA Cleansing Gel: Used twice daily (AM and PM) to cleanse the skin and target discoloration.
  Hydrating B5 Gel: Applied throughout the day to hydrate the skin. Brightening UV Defense Sunscreen: Used throughout the day.
  Interventions: Other: Pigment Balancing Peel; Other: Discoloration Defense Serum; Other: LHA Cleansing Gel; Other: Hydrating B5 Gel; Other: Daily Brightening Sunscreen

INTERVENTIONS:
Other: Pigment Balancing Peel — Chemical Peel
Other: Discoloration Defense Serum — Dark spot correcting serum
Other: LHA Cleansing Gel — exfoliating gel facial cleanser
Other: Hydrating B5 Gel — Vitamin B5 serum with hyaluronic acid
Other: Daily Brightening Sunscreen — daily moisturizing sunscreen SPF 30

SUMMARY:
This is a single-center, prospective, non-blinded, non-randomized 12 week clinical study to evaluate the efficacy of a SkinCeuticals comprehensive skin care regimen in the reduction of post inflammatory hyperpigmentation (PIH) in skin of color patients. The comprehensive regimen features the Pigment Balancing Peel which combines glycolic acid, lactic acid, kojic acid, vitamin C, and emblica into a treatment that may improve skin discoloration. Participants will supplement the Pigment Balancing Peel with a 11 week regimen that includes the Hydrating B5 Gel, Discoloration Defense, LHA Cleansing Gel, and Brightening UV Defense sunscreen.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ages 18+.
* Clinical diagnosis of Post Inflammatory Hyperpigmentation
* Non-Caucasian
* Fitzpatrick skin types IV-VI
* Available and willing to comply with study instructions and attend all study visits.
* Able and willing to provide written and verbal informed consent.

Exclusion Criteria:

* Subject has any skin pathology or condition that could interfere with the evaluation of the test products or requires the use of interfering topical or systemic therapy.
* Caucasian/ Non-Hispanic
* Subject has any condition which, in the investigator's opinion, would make it unsafe for the subject to participate in this research study.
* Pregnant, lactating, or is planning to become pregnant during the study.
* Subject is currently enrolled in an investigational drug or device study.
* Subject has received an investigational drug or has been treated with an investigational device within 30 days prior to the initiation of treatment (baseline).
* Study participant has facial hair that could interfere with the study assessments in the opinion of the investigator.
* Study participant is unable to communicate or cooperate with the investigator due to language problems, poor mental development, or impaired cerebral function.
* Subject has known hypersensitivity or previous allergic reaction to any of the active or inactive components of the test articles.
* Subject has the need or plans to be exposed to artificial tanning devices or excessive sunlight during the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-02-28 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline to week 12 of patient satisfaction in improvement of post-inflammatory hyperpigmentation | From enrollment to end of treatment at 12 weeks
  Change in the patient satisfaction with their physical appearance following use of SkinCeuticals regimen to improve post inflammatory hyperpigmentation, using the FACE-Q Satisfaction (scores range from 0 (lowest) to 100 (highest)), at week 12 compared to baseline.

SECONDARY OUTCOMES:
Change in DLQI at baseline vs week 12 | From enrollment to end of treatment at 12 weeks
  Change in the DLQI (ranges from 0 (no impact on quality of life) to 30 (maximum impairment)) following use of Pigment Balancing Peel, Hydrating B5 Gel, Discoloration Defense, LHA Cleanser Gel and Brightening Sunscreen, at baseline vs week 12.
Change in the melanin and erythema index at baseline, week 6, and week 12 | From enrollment to end of treatment at 12 weeks
  Change in the melanin (0-999) and erythema (0-999) index measured by the Delfin SkinColorCatch at baseline, week 6 and week 12. (0 is lightest and 100 is darkest)
Patient expectations utilizing FACE-Q Expectations Scale | From enrollment to end of treatment at 12 weeks
  To assess patient expectations regarding the impact of treatment on their lives utilizing FACE-Q Expectations Scale (scores range from 0 (lowest) to 100 (highest)), as completed by the patient at baseline visit.
Change in psychosocial factors utilizing the FACE-Q Social Function Scale following treatment at baseline vs week 12 | From enrollment to end of treatment at 12 weeks
  To evaluate changes in psychosocial factors following aesthetic treatment, utilizing FACE-Q Social Function Scale (scores range from 0 (lowest) to 100 (highest)) as completed by the patient at baseline vs week 12.
Change in psychosocial factors utilizing the FACE-Q Psychological Function Scale following treatment at baseline vs week 12 | From enrollment to end of treatment at 12 weeks
  To evaluate changes in psychosocial factors following aesthetic treatment, utilizing FACE-Q Psychological Function Scale (scores range from 0 (lowest) to 100 (highest)) as completed by the patient at baseline vs week 12.
Patient satisfaction with treatment using FACE-Q outcome scale at week 12 | From enrollment to end of treatment at 12 weeks
  To assess patient satisfaction with treatment using the FACE-Q Outcome Satisfaction Scale, (scores range from 0 (lowest) to 100 (highest)) as completed by the patient at week 12

CONTACTS AND LOCATIONS:
Overall Officials: Jared Jagdeo, MD MS, Principal Investigator — SUNY Downstate Health Sciences University Department of Dermatology
Locations (1):
- New York Harbor VA Brooklyn Campus, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided